CLINICAL TRIAL: NCT02072213
Title: A Randomized, Open-label, Single-dose, Four-sequence, Four -Period Crossover Study to Investigate The Pharmacokinetics of GL2702 GLARS-NF1 and Omix Ocas® in Healthy Male Volunteers
Brief Title: A PK Study GL2702 GLARS-NF1 and Omix Ocas® in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GL Pharm Tech Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GL2702-103
Record Dates: First submitted 2014-02-24; First posted 2014-02-26 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2014-02

CONDITIONS: Healthy
Keywords: Tamsulosin,controlled release formulation
MeSH Terms: interventions — Tamsulosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- GL2702 GLARS-NF1 , fasted (Experimental): Tamsulsoin 0.4mg
  Interventions: Drug: GL2702 GLARS-NF1
- Omix Ocas® , fasted (Active Comparator): Tamsulsoin 0.4mg
  Interventions: Drug: Omix Ocas
- GL2702 GLARS-NF1, after meal (Experimental): Tamsulsoin 0.4mg
  Interventions: Drug: GL2702 GLARS-NF1
- Omix Ocas®, after meal (Active Comparator): Tamsulsoin 0.4mg
  Interventions: Drug: Omix Ocas

INTERVENTIONS:
Drug: GL2702 GLARS-NF1 — 0.4mg once a day
  Other Names: Tamsulosin
  Arms: GL2702 GLARS-NF1 , fasted; GL2702 GLARS-NF1, after meal
Drug: Omix Ocas — 0.4mg once a day
  Other Names: Tamsulosin
  Arms: Omix Ocas® , fasted; Omix Ocas®, after meal

SUMMARY:
Study to Investigate The Pharmacokinetics of GL2702 GLARS-NF1 and Omix Ocas® in Healthy Male Volunteers

DETAILED DESCRIPTION:
GL2702 GLARS-NF1 tablet is controlled released formulation which is invented by GL Pharm Tech Corp.

ELIGIBILITY:
Inclusion Criteria:

* 20~45 years old, Healthy Adult Male Subject
* Body Weight ≥ 50kg and Ideal Body Weight ≤ ±20%

Exclusion Criteria:

* ALT or AST > 1.25 times (Upper Normal Range)
* Total Bilirubin > 1.5 times (Upper Normal Range)
* CPK > 2 times (Upper Normal Range)
* BUN or Creatinine > Normal Range
* Systolic BP > 160mmHg or < 80mmHg, Diastolic BP > 100mmHg or < 50mmHg

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Cmax | 48 hours
  Pharmacokinetic parameter of tamsulosin 0.4mg
AUClast | 48 hours
  Pharmacokinetic parameter of Tamsulosin 0.4mg

SECONDARY OUTCOMES:
Tmax | 48 hours
  Pharmacokinetic parameter of Tamsulosin 0.4 mg
t1/2 | 48 hours
  Pharmacokinetic parameter of Tamsulosin 0.4 mg
Vz/F | 48 hours
  Pharmacokinetic parameter of Tamsulosin 0.4 mg
CL/F | 48 hours
  Pharmacokinetic parameter of Tamsulosin 0.4 mg

CONTACTS AND LOCATIONS:
Overall Officials: Min-Gul Kim, MD, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, Jeollabukdo, South Korea